CLINICAL TRIAL: NCT03157856
Title: Assessment of a New Fluorescence Imaging Technique Using Biopsies From Prostate Resection
Acronym: Bio-Prost
Status: Terminated | Type: Observational
Why Stopped: Results obtained on the first 8 patients shown an expected glandular membrane specific labeling associated with non-specific labeling of fibro-muscular tissue.
Sponsor: University Hospital, Grenoble (Other)
Collaborators: TIMC-IMAG (Other); Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor
Other Study IDs: 38RC17.019
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Cancer Prostate
Keywords: Fluorescence imaging technique; Biopsies from resected prostate; Medical device
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: fluorescence assessment: Medical device: Use of the FEMTO-ST institute medical device to detect prostatic and non prostatic tissue.
  Interventions: Other: Fluorescence assessment

INTERVENTIONS:
Other: Fluorescence assessment — All subjects of the study are going to have a radical prostatectomy. The FEMTO-ST medical device is used on 3 fresh biopsies (2 healthy and 1 malignant) which will be prelevated from the resected prostate in order to determine the prostatic or non-prostatic nature of tissue.

SUMMARY:
In this study, we aim to evaluate the feasibility of anti-PSMA labelling to detect post-operative prostatic tissues by two ex vivo fluorescence techniques. We will evaluate the feasibility and detection of anti-PSMA labelling by:

1. / the FEMTO-ST institute medical device,
2. / the confocal microscope that will be used to measure fluorescence spectra of biological samples.

DETAILED DESCRIPTION:
For this protocol, 12 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* male patient over 18 years old
* patient with indication for radical prostatectomy
* patient with a rectal palpable nodule or targeted MRI positive biopsies or with at least 4 positive biopsies in a hemi-prostate.

  * patient affiliated to French social security system or equivalent
  * patient who have signed a non-opposition form

Exclusion Criteria:

* patient with contraindication to radical prostatectomy
* patient with remedial prostatectomy
* patient with normal preoperative MRI or with absence of tumoral area
* patient with history of hormonal therapy
* person deprived of freedom by judicial or administrative decision
* person under legal protection
* person hospitalized for psychiatric care.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with indication for radical prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2018-10-07 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Comparison of the fluorescence obtained using the FEMTO-ST device and the confocal microscope of anti-PSMA marked fresh prostate biopsies, for prostatic and non-prostatic tissue, as identified by anatomo-pathology (gold standard). | 14 months
  Fluorescence measurements obtained using the FEMTO-ST medical device and the confocal microscope.

SECONDARY OUTCOMES:
Comparison of the fluorescence obtained using the FEMTO-ST device and the confocal microscope of anti-PSMA marked fresh prostate biopsies, for cancerous and non-cancerous tissue, as identified by anatomo-pathology (gold standard). | 14 months
  Fluorescence measurements obtained using the FEMTO-ST medical device and the confocal microscope.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Luc Descotes, MD, PhD, Principal Investigator — Grenoble Alpes University Hospital
Locations (2):
- France (2):
  - Grenoble Alpes University Hospital - Urology department, Grenoble
  - Grenoble Alpes University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: No